CLINICAL TRIAL: NCT03608657
Title: Observational Study Evaluating the Real-World Effectiveness, Safety and Tolerability of Treatment With Apremilast in Psoriatic Arthritis Patients Followed in Canadian Routine Care (APPRAISE)
Brief Title: Study to Evaluate the Real-World Effectiveness, Safety and Tolerability of Treatment With Apremilast in Psoriatic Arthritis Patients Followed in Canadian Routine Care (APPRAISE)
Acronym: APPRAISE
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSA-011; U1111-1214-0693 (Other: UTN)
Record Dates: First submitted 2018-05-30; First posted 2018-08-01 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Arthritis, Psoriatic
Keywords: Psoriatic Arthritis; Canada; CC-10004; Apremilast; APPRAISE; Safety; Non-interventional; Observation; DMARDs
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — apremilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Psoriatic Arthritis patients treated with Apremilast: Active PsA as per the CASPAR criteria, based on the investigator's clinical judgement with access to commercially available Otezla
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast
  Other Names: Otezla

SUMMARY:
This will be a Canadian observational study utilizing a prospective cohort design. Patients with active psoriatic arthritis (PsA) for whom the treating physician has decided, prior to and independently of enrollment in the study, to initiate treatment with Otezla® will be considered for participation in the study.

Patients will be enrolled from the practices of predominantly community rheumatologists and will be followed for 12 months from the time of initiation of treatment with Otezla® In line with the observational nature of the study, there will be no protocol imposed tests or assessments. However, recommended follow up visits will be at 4, 8 and 12 months. In addition, patients may be asked to voluntarily complete self-administered questionnaires.

The 24-month assessment will be aimed to determine whether or not treatment with Otezla® has been maintained, and if not, to ascertain the reason for discontinuation and what new treatment was initiated following discontinuation of Otezla®

ELIGIBILITY:
Inclusion Criteria:

* Active psoriatic arthritis (PsA) as per the Classification criteria for Psoriatic Arthritis (CASPAR) criteria, based on the investigator's clinical judgement.
* Adult patients (≥18 years of age) with PsA
* Prescribing physician has decided to initiate treatment with Otezla®, and this decision was prior to and independent of patient enrollment in the study.
* Access to commercially available Otezla®

Exclusion Criteria:

* Patients who are pregnant, breastfeeding, or who are planning on becoming pregnant during the course of the study
* Participation in Investigational Clinical Trial within the last 60 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with active PsA and access to commercial Otezla® who are under the care of a Canadian rheumatologist.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
The rate of achieving Low Disease Activity (LDA) | Up to approximately 1 year
  Is defined as Clinical Disease Activity Index for Psoriatic Arthritis (cDAPSA) < 14. cDAPSA is calculated as the sum of TJC - 68, SJC - 66, PtGA (10-cm VAS) and Pain (10-cm VAS).

SECONDARY OUTCOMES:
The rate of achieving Low Disease Activity (LDA) | Up to approximately 8 months
  Is defined as Clinical Disease Activity Index for Psoriatic Arthritis (cDAPSA) < 14. cDAPSA is calculated as the sum of TJC - 68, SJC - 66, PtGA (10-cm VAS) and Pain (10-cm VAS).
Tender Joint Count (TJC) | Up to Approximately 1 year
  Based on 68/66 joints to determine joint pain/tenderness and joint swelling, as conducted during the physical examination and per the practices of the treating physician
Swollen Joint Count (SJC) | Up to Approximately 1 year
  Based on 68/66 joints to determine joint pain/tenderness and joint swelling, as conducted during the physical examination and per the practices of the treating physician
Assessment of Enthesitis (Leeds Enthesitis Index (LEI) | Up to Approximately 1 year
  This is completed by the treating physician and assesses tenderness at six (6) sites, specifically two (2) lateral at the following: epicondyles of the humerus, medial condyles of the femur and the insertion of the Achilles tendon. The LEI is scored between 0 and 6. Resolution versus improvement versus no change versus worsening of enthesitis since the last available assessment
Assessment of Dactylitis (Leeds Dactylitis Index) | Up to approximately 1 year
  Resolution versus improvement versus no change versus worsening of dactylitis since the last available assessment
Assessment of Body Surface Area (BSA) | Up to approximately 1 year
  height (cm) x weight (kg)/3600)½
Health Assessment Questionnaire Disability Index (HAQ-DI) | Up to approximately 1 year
  This is a self-administered questionnaire measuring the patient's functional ability during the last week. It consists of 20 items converging to 8 scales measuring dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. The patients rate each activity as 0 = without any difficulty, 1 = some difficulty, 2 = much difficulty and 4 = unable. The final score ranges from 0 to 3 with higher scores indicating more disability.
Physician global assessment of disease activity (MDGA) | Up to approximately 1 year
  This is a 100-mm visual analog scale (VAS) with 0 indicating lowest disease and 100 highest disease activities
Patient global assessment of disease activity (PtGA) | Up to approximately 1 year
  This is a 100-mm VAS with 0 indicating lowest disease and 100 highest disease activity
Treatment Satisfaction Questionnaire for Medication (TSQM) | Up to approximately 1 year
  This is a 14-item questionnaire evaluating patient satisfaction in terms of the following: effectiveness, side effects, convenience, and global satisfaction
Patient subjective assessment of Pain using a 100mm VAS | Up to approximately 1 year
  Patient subjective assessment of Pain using a 100mm VAS
Psoriatic Arthritis (WPAI:PsA) | Up to approximately 1 year
  A 6-item questionnaire assessing the effect of PsA on the patient's ability to work and perform daily activities. It assesses presenteeism, absenteeism, productivity and activity impairment
Medical Outcomes Study Short- Form 36 (SF-36) | Up to approximately 1 year
  A generic quality of life index that is comprised of 36 items converging to eight (8) domains: Vitality, Physical Functioning, Bodily Pain, General Health Perception, Physical Role Functioning, Emotional Role Functioning, Social Role Functioning, and Mental Health
Patient-reported adherence with PsA treatment from the last visit. | Up to approximately 1 year
  An optional weekly take-home diary will be offered to patients; this diary will aid in documenting how many doses (if any) of PsA treatment were missed, and the reason(s) why.
Proportion of patients in Patient Acceptable Symptom State (PASS) | Up to approximately 1 year
  A single question phrased as "If you were to remain for the next few months as you were during the last week, would this be acceptable or unacceptable to you?" with a binary (Yes or No) response
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  Number of subjects with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (19):
- Canada (19):
  - The Waterside Clinic, Barrie
  - The Arthritis and Osteoporosis Centre, Burlington
  - Adachi Medicine Professional Corporation, Hamilton
  - Credit Valley Rheumatology, Mississauga
  - Institut de Recherche en Rhumatologie de Montréal, Montreal
  - Applied Medical Informatics Research Inc. (A.M.I.R.), Montreal
  - Brent Appleton Clinic New Westminster, New Westminster
  - Dr. A. M. Jaroszynska Rheumatology and Osteoporosis Clinic, Oakville
  - Drs M&W Teo, Penticton
  - Groupe de recherche en maladies osseuses Inc., Québec
  - Centre de Rhumatologie de l'Est du Quebec, Rimouski
  - Polmed Research Inc., Saskatoon
  - Clinique Jacques Cartier, Sherbrooke
  - St. Clare's Mercy Hospital, St. John's
  - Dr. Juris Lazovskis Incorporated, Sydney
  - Toronto Western Hospital, University Health Network, Toronto
  - Arthur Karasik Medicine Professional Inc., Toronto
  - Dr. Jonathan D. Chan Inc., Vancouver
  - Dr. Sabeen Anwar Medicine Professional Corporation, Windsor

REFERENCES:
- [Derived] Chandran V, Bessette L, Thorne C, Sheriff M, Rahman P, Gladman DD, Anwar S, Jelley J, Gaudreau AJ, Chohan M, Sampalis JS. Use of Apremilast to Achieve Psoriatic Arthritis Treatment Goals and Satisfaction at 1 Year in the Canadian Real-World APPRAISE Study. Rheumatol Ther. 2024 Apr;11(2):443-455. doi: 10.1007/s40744-024-00641-w. Epub 2024 Feb 28. PMID 38416391
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Expanded Access for CC-10004 — https://clinicaltrials.gov/ct2/show/NCT03608657?term=CC-10004-PSA-011&rank=1